CLINICAL TRIAL: NCT04564378
Title: Association Between Fuchs' Endothelial Corneal Dystrophy Severity and Estrogen Exposure
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Sangita Patel, Assistant Professor, State University of New York at Buffalo
Other Study IDs: STUDY00002020
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Fuchs Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild Fuchs Dystrophy
  Interventions: Other: This is an observational study. There is no therapeutic intervention.
- Severe Fuchs Dystrophy
  Interventions: Other: This is an observational study. There is no therapeutic intervention.

INTERVENTIONS:
Other: This is an observational study. There is no therapeutic intervention. — This is an observational study. There is no therapeutic intervention.

SUMMARY:
This study is being done to discover if there is a link between estrogen exposure and the severity of Fuchs Endothelial Corneal Disease. We are trying to understand if the decrease in estrogen levels in post-menopausal women may be a reason why FECD is seen more often in women than men.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with FECD grade 1-2/7 (mild) or 5-6/7 (severe) in one or both eyes
2. Age ≥ 55
3. Phakic and pseudophakic individuals will be included. Pseudophakic patients must have evidence of routine cataract surgery (posterior chamber intraocular lens in-the-bag without clinical evidence of damage to any intraocular structures).

Exclusion Criteria:

1. Females are excluded if not post-menopause.
2. Pseudophakic patients with a history of complex cataract surgery or other intraocular surgery (e.g. have an anterior chamber lens, sulcus lens, or poorly positioned posterior chamber lens, aphakia, iris damage, glaucoma surgery) will be excluded due to risk of iatrogenic damage to the corneal endothelium.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with mild or severe Fuchs Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Association Between Fuchs endothelial Corneal Dystophy Severity and Estrogen Exposure | 5 years
  Difference in measures of estriadiol exposure between individuals with mild vs. severe FECD

CONTACTS AND LOCATIONS:
Overall Officials: Sagita Patel, Principal Investigator — The Ross Eye Institute
Locations (1):
- The Ira G. Ross Eye Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No